CLINICAL TRIAL: NCT03947034
Title: Monitoring the Hyperammonaemia:TOXicity of Drugs (AmmoTOX)
Acronym: AmmoTOX
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Principal Investigator, Joe Elie Salem, Assistant director, clinical investigation center Paris Est, Groupe Hospitalier Pitie-Salpetriere
Other Study IDs: CIC1421-19-09
Record Dates: First submitted 2019-05-09; First posted 2019-05-13 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Hyperammonemia; Metabolic Disease; Adverse Drug Event; Drug Toxicity
MeSH Terms: conditions — Hyperammonemia; Metabolic Diseases; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Metabolic toxicity induced by drugs and chemotherapies: Case reported in the World Health Organization (WHO) of metabolic toxicities(such as hyperammonemia) of patient treated by a drug, with a chronology compatible with the drug toxicity
  Interventions: Drug: Drugs inducing hyperammonemia

INTERVENTIONS:
Drug: Drugs inducing hyperammonemia — Drugs susceptible to induce metabolic toxicities such as hyperammonemia

SUMMARY:
Several drugs and chemotherapies seem to have an impact on the metabolic system. This study investigates reports of metabolic toxicities such as hyperammonemia, including the International classification of disease ICD-10 for treatments in the World Health Organization (WHO) global Individual Case Safety Report (ICSR) database (VigiBase).

DETAILED DESCRIPTION:
Several drugs and chemotherapies seem to have an impact on the metabolic system and are responsible of a wide range of metabolical side effects such as hyperammonemia. Those are poorly described, due to the modification of the pharmacopeia, and the recent recognition of several of these adverse events. This study investigates the main characteristics of patients affected by metabolic side effects imputed to drugs in particular hyperammonemia. A causality assessment according to the WHO-UMC (World Health Organization - Uppsala Monitoring Center) is systematically applied.

ELIGIBILITY:
Inclusion Criteria:

* Case reported in the WHO's pharmacovigilance database till 01/05/2019

Exclusion Criteria:

* Chronology not compatible between the drug and the toxicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with a drug that could be reported in the WHO's pharmacovigilance database
Sampling Method: Non-Probability Sample
Enrollment: 2700 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Metabolic toxicities (such as hyperammnemia) of drugs Identification and report of cases of metabolic toxicities associated with drugs. | to 01/05/2019
  Case reported in the World Health Organization (WHO) database of individual safety case reports

SECONDARY OUTCOMES:
Causality assessment of reported metabolic toxicities events according to the WHO system | to 01/05/2019
  Case reported in the World Health Organization (WHO) database of individual safety case reports
Description of the type of metabolic toxicity depending on the category of drug | to 01/05/2019
  Case reported in the World Health Organization (WHO) database of individual safety case reports
Description of the other immune related adverse events concomitant to the metabolic toxicity induced by drugs | to 01/05/2019
  Case reported in the World Health Organization (WHO) database of individual safety case reports
Description of the duration of treatment when the toxicity happens (role of cumulative dose) | to 01/05/2019
  Case reported in the World Health Organization (WHO) database of individual safety case reports
Description of the drug-drug interactions associated with adverse events | to 01/05/2019
  Case reported in the World Health Organization (WHO) database of individual safety case reports
Description of the pathologies (cancer) for which the incriminated drugs have been prescribed | to 01/05/2019
  Case reported in the World Health Organization (WHO) database of individual safety case reports
Description of the population of patients having hematological toxicity adverse event | to 01/05/2019
  Case reported in the World Health Organization (WHO) database of individual safety case reports

CONTACTS AND LOCATIONS:
Locations (1):
- AP-HP, Pitié-Salpêtrière Hospital, Department of Pharmacology, CIC-1421, Pharmacovigilance Unit, INSERM, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided